CLINICAL TRIAL: NCT00878423
Title: A Phase I Open-label Dose Escalation Study of AT13387 in Patients With Metastatic Solid Tumors
Brief Title: Study to Assess the Safety of Escalating Doses of AT13387 in Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AT13387/0001
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Solid Tumors
Keywords: HSP90; Metastatic solid tumor including lymphoma which are; refractory to standard therapy
MeSH Terms: interventions — (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AT13387 — Two dosing schedules will be evaluated; twice or once weekly dosing, on three weeks out of four. The starting dose for the once weekly schedule was 10mg/m2/dose, given as one hour intravenous (IV) infusions on Days 1, 4, 8, 11, 15 and 18 of a twenty-eight day cycle. The starting dose for the twice weekly schedule, given as one hour intravenous (IV) infusions on Days 1, 8 and 15 of a twenty-eight day cycle, will be 150mg/m2/dose
Drug: AT13387 — Intravenous infusion over one hour on days 1, 4, 8, 11, 15 and 18, every four weeks or intravenous infusion over one hour on days 1, 8 and 15, every four weeks . Treatment may be continued indefinitively in the presence of clinical benefit

SUMMARY:
AT13387/0001 is a dose-finding study of an experimental anticancer agent. In accordance with the protocol increasing doses of AT13387 are given to patients with advanced cancer who do not have alternative treatment options. The preferred dose of AT13387 will be identified according to the side effects experienced at different dose levels.

DETAILED DESCRIPTION:
Increasing doses of AT13387 will be administered to groups of 3 to 6 patients at each dose level. The pharmacokinetic profile of AT13387 following a one hour intravenous infusion will be determined and the effect of AT13387 on predefined biomarkers in blood plasma and circulating white blood cells will be established. Patients will be closely monitored for the development of side effects which would preclude further dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent.
* Age 18 years or older.
* Histological or cytological evidence of a metastatic solid tumor including lymphoma, which is refractory to standard therapy. The following tumor types are of particular interest as they may be more likely to respond to HSP90 inhibition and all efforts should be made to recruit patients into the study with these diagnoses. Only patients with these diagnoses and others thought to be responsive to HSP90 inhibitors are to be enrolled following the identification of MTD.

  * Metastatic breast cancer which is HER2 positive either by FISH or 3+ immunohistochemistry staining,
  * Adenocarcinoma of the prostate which is refractory to treatment with androgen depletion,
  * Metastatic melanoma,
  * Stage IIIb or IV NSCLC,
  * SCLC,
  * High grade gliomas (patients must have been on a stable dose of corticosteroids for at least one week prior to treatment with AT13387 and have not experienced neurological deterioration during this period),
  * GIST.
* ECOG performance status ≤ 2.
* Adequate marrow function as defined by:

  * Hemoglobin > 9 g/dL,
  * Neutrophils > 1.4 x 10^9/L,
  * Platelets ≥ 100 x 10^9/L.
* Negative serum or urine pregnancy test or evidence of surgical sterility or evidence of post-menopausal status. Post-menopausal status is defined as any of the following: natural menopause with menses >1 year ago; radiation induced oophorectomy with last menses >1 year ago; chemotherapy-induced menopause with 1 year interval since last menses.

Exclusion Criteria:

* Be pregnant or lactating (women of childbearing potential must have a negative pregnancy test within 7 days prior to enrolment). Male and female patients of childbearing potential must use appropriate birth control (barrier methods, oral contraceptives and/or intrauterine devices) during the entire duration of the study, or the patient must be surgically sterile (with documentation in the patient's medical records).
* Ongoing central nervous system metastases in patients with an extracranial primary tumor (unless the patient's neurological signs or symptoms have been stable during the preceding three months and the patient has not received corticosteroid treatment for four weeks prior to study entry).
* Inadequate liver function as demonstrated by serum bilirubin > 2.5 times the upper limits of reference range (ULRR) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or alkaline phosphatase (ALP) ≥ 2.5 times the ULRR (unless due to the presence of liver metastases when ALT and/or AST may be up to five times the upper limits of reference range). Patients with an isolated increase in ALP ≤ 5 times ULRR in the absence of liver metastases but with known bone metastases are eligible for the study.
* Left ventricular ejection fraction <50% on echocardiography or MUGA scan.
* Moderate or severe renal impairment defined as serum creatinine > 1.5 ULRR or > + proteinuria on two occasions no less than 24 hours apart.
* Previous treatment with a HSP90 inhibitor.
* Anticancer therapies that have not been completed at least 28 days prior to treatment with AT13387 (other than surgery or treatment with a protein kinase inhibitor which must have been completed no less than one week prior to treatment with AT13387).
* Incomplete recovery from previous radiotherapy or surgery other than residual cutaneous effects or stable < Grade 2 gastrointestinal toxicity.
* History of an ischemic cardiac event, myocardial infarction or unstable cardiac disease within 3 months of study entry.
* QTc > 460 ms according to the Fridericia's correction.
* Previous malignancy, except for non-basal-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix, unless the tumor was treated with curative intent more than 2 years prior to study entry.
* Any evidence of severe or uncontrolled systemic conditions (e.g., systemic infection) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
* Prior history of infection with human immunodeficiency virus (HIV), known active hepatitis B or C viruses - screening for viral infections is not required for entry to this study.
* Chronic treatment with known CYP450 inducers e.g. phenytoin, within four weeks of receiving treatment with AT13387 (see Appendix D for list) other than Dexamethasone in patients with glioma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-05; Primary Completion 2013-05 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The identification of the maximum tolerated dose for twice or once weekly dosing, on three weeks out of four | 12 months

SECONDARY OUTCOMES:
Pharmacokinetic profile, Safety and tolerability of maximum tolerated dose, pharmacodynamic effect, identify dose limiting toxicities | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts